CLINICAL TRIAL: NCT06784245
Title: Effectiveness of Synchronous Telerehabilitation Versus Face-To-Face Physical Therapy on Physical Fitness, Functional Status, and Quality of Life in Frail Older Adults
Brief Title: Telerehabilitation on Physical Fitness, Functional Status, and Quality of Life in Frail Older Adults
Acronym: Teleactivate 3
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Marina Alvarado (Other)
Responsible Party: Sponsor-Investigator, Marina Alvarado, PhD, Universidad Catolica Silva Henriquez
Organization: Universidad Catolica Silva Henriquez (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: F. iniciacion n°11240532; 11240532 (Other Grant/Funding Number: Agencia Nacional de Investigación y Desarrollo (ANID))
Record Dates: First submitted 2025-01-14; First posted 2025-01-20 (Actual); Last update posted 2025-02-03 (Actual); Status verified 2025-01

CONDITIONS: Frailty At Older Adults
Keywords: Older person; Fragility; Telerehabilitation; Physical fitness; Functional status; Quality of life
MeSH Terms: interventions — Telerehabilitation

STUDY DESIGN:
Intervention Model Description: Synchronous telerehabilitation program (STR group) During the exercise session, the participants turns on the tablet PC, watches the instructor perform the exercise, and follows the instructor's movements. For the instructor to observe the correct movements of the participants, the resistance and balance exercises are performed in the frontal and sagittal planes. During each session, a technical stuff will supervise up to four or five participants exercising remotely at home, using a real-time videoconferencing app (Zoom®, CA, USA). The videoconference session will be projected on a television screen located in an older adult's care center. Once the technical stuff has been assigned participants, their supervision will not be interchangeable. Participants will be able to see and talk to both, the healthcare professional and other participants. The older adults, from their homes, will complete 1-hour sessions, twice a week for 12 weeks.
Who Masked: Outcomes Assessor
Masking Description: This study has been designed as a blinded (assessor and statistician), parallel group, randomized controlled trial (RCT)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Synchronous telerehabilitation program (STR Group) (Experimental): During each session, a technical staff member will supervise up to four or five participants who are exercising remotely at home using a real-time videoconferencing app (Zoom®, CA, USA). The videoconference session will be projected on a television screen located in an older adult's care centre. Participants will be able to see and talk to the healthcare professional and other participants. The older adults, from their homes, will complete 1-hour sessions twice a week for 12 weeks.
  Interventions: Behavioral: TeleActivate
- Face-to-face physical therapy program (FPT Group) (Active Comparator): The face-to-face exercise sessions will take place in a senior centre for older person, lasting 40-60 min, twice a week for 12 weeks.
  Interventions: Behavioral: TeleActivate

INTERVENTIONS:
Behavioral: TeleActivate — Each session will consist of a warm-up activity (5-10 min), main exercise activity (30-40 min), and cool-down activity (5-10 min) following the guidelines of multicomponent exercise program Vivifrail. Exercise intensity will be controlled based on the Rating of Perceived Exertion (RPE) on the Borg scale and heart rate measured with a smartwatch before, during, and after each exercise session according to the guidelines of the American College of Sports Medicine (ACSM), as explained below. The warm-up and cool-down activities will include stretching and walking in place (9≤RPE≤10 and 40<55% maximum Heart rate (HRmax). While the main exercise activity will consist of strength, resistance exercise, cardiovascular exercises, and balance exercises (to avoid falls) performed using dumbbells, colour-coded resistance bands (Thera-Band; Hygenic Corp.) and a chair (11<RPE≤15 and 55<70 HRmax).
  Other Names: Telerehabilitation

SUMMARY:
The goal of this randomized controlled trial (RCT) is to analyze whether the effectiveness of a synchronous telerehabilitation program is better than a face-to-face physical therapy program in improving the physical fitness, functional status, and quality of life in frail male and female volunteers aged 60 years or older living in the community and haven frailty according to the modified Fried phenotype scale. The main research questions are: 1) Is a synchronous telerehabilitation program effective in improving the physical fitness, functional status and quality of life of frail older people?; 2) Is a synchronous telerehabilitation program more effective in improving the physical fitness, functional status and quality of life, compared to face-to-face physical therapy program, in frail older adults? In synchronous telerehabilitation program group, a healthcare professional will supervise up to four or five participants remotely exercising at home during each session, using a real-time videoconferencing app. Participants will be able to see and talk to both the health professional and the other participants. The exercise program will consist of 1-hour sessions carried out twice a week for 12 weeks. In the face-to-face physical therapy group, the exercise sessions will take place in a older person care center, which will also last 1 hour twice a week for 12 weeks. Regardless of the group, exercise sessions will include a mixture of cardiovascular, balance, strength, flexibility, and gait exercises.

DETAILED DESCRIPTION:
Background A promising solution to solve the barriers to practice physical activity in frailty older adults (OAs) is the incorporation of a synchronous telerehabilitation program. Mobile technologies are emerging tools that have the potential to facilitate health care, reduce distance barriers, time, and cost, that limits accessibility to face-to-face physical therapy program, facilitates access to opportunities and reduces healthcare gaps. Nevertheless, there is little evidence of its effectiveness as a therapeutic strategy and more rigorous studies are suggested. To date, a few studies in Chile have used mobile apps to support the treatment of OAs regarding physical fitness and functional status and there are no studies that have analyzed the effects of synchronous telerehabilitation in OAs.

General objective To analyze whether the effectiveness of a synchronous telerehabilitation program is better than a face-to-face physical therapy program in improving the physical fitness and functional status, and quality of life in frail older adults.

Methodology A blinded, parallel group, randomized controlled trial (RCT), Adults ≥60 years old from Los Ángeles, Chile, will be recruited. The inclusion criteria will be: (i) both sexes aged ≥60 years, (ii) community-dwelling older adults, (iii) Older adults having frailty according to the modified Fried phenotype scale (ref), (iv) ability to stand up and walk ≥10 meters without assistance technique, (v) Abbreviated Mini Mental State (MMSE) >13 points, (vi) without medical contraindication for physical exercise. Exclusion criteria includes those older adults presenting fractures and recent acute myocardial infarction, associated cardiovascular pathology, severe acute respiratory failure, high blood pressure, uncontrolled diabetes mellitus, limitations following instructions as well as people participating in other exercise program during the project. The sample size was calculated a priori using G*Power 3.1.9.7., the total of subjects required is 52. (26 in each group) considering α=0.05, 1-β=0.8 and effect size (ES)=0.8. Having in consideration the possibility of abandonment, 6 subjects were added (total n=58; n=29 in each group). Participants who meet the participation criteria will be randomized using a computer-generated sequence and concealed allocation to one of the following two groups:(1) STR Group who performed synchronous telerehabilitation, or (2) the FPT Group who performed face-to-face physical therapy.

Procedures:

Physical fitness, functional status, and quality of life will be assessed face-to-face 1 week prior to initiating the intervention in both groups.

Additionally, at that time, STR group participants will be provided with a tablet and home exercise equipment (exercise mats, resistance bands, cones, and dumbbells). If exercise materials are lost or damaged, they will be replaced. A home visit will be made to identify barriers to exercise and determine the right place to carry out the synchronous telerehabilitation sessions. Written and verbal instructions will be given outlining the simple steps necessary to connect to an online meeting and facilitating participation in the synchronous telerehabilitation program as well as on the proper use of the home exercise equipment. At the beginning of the interventions, all participants will be given a hydration kit (cotton towel and a water bottle) a smartwatch (Fitbit® Inspire 2, by Google, California, USA) to measure continuous heart rate monitoring during exercise sessions to maintain exercise intensity, and pedometer (OMRON® HJ-321, Kyoto, Japan) to record the number of daily steps each participant takes.

The home exercise equipment and technological equipment (tablet, pedometer, and smartwatch) will be delivered to the participants through the signing of a loan agreement and will be returned to the responsible researcher once the data collection is finished. If the technological equipment presents a factory defect during the execution of the study, the 12-month manufacturer's guarantee will be used. During the intervention period, nutrition guidance and exercise education will be provided to all participants once every 4 weeks. Throughout the 12-week intervention period, the participants will be encouraged to maintain the same physical activity levels and calorie intake as before participating in the study. During educational sessions, the investigators will ask participants to report to session staff any changes in their physical activity levels or nutritional intake during the intervention period. A postintervention assessment will be performed after the last week of the 12-week program. All data collection will be carried out in a face-to-face meeting with older adults at a care center. Technical stuff will be trained, which will guarantee an unbiassed procedure. Measurements will be obtained individually, in a place with optimal conditions of privacy, temperature and humidity. Evaluations will be acquired by healthcare professionals; the person evaluating will be different to the one performing the interventions.

Interventions:

Synchronous telerehabilitation program (STR group) During the exercise session, the participants turns on the tablet PC, watches the instructor perform the exercise, and follows the instructor's movements. For the instructor to observe the correct movements of the participants, the resistance and balance exercises are performed in the frontal and sagittal planes. During each session, a technical stuff will supervise up to four or five participants exercising remotely at home, using a real-time videoconferencing app (Zoom®, CA, USA). The videoconference session will be projected on a television screen located in an older adult's care center. Once the technical stuff has been assigned participants, their supervision will not be interchangeable. Participants will be able to see and talk to both, the healthcare professional and other participants. The older adults, from their homes, will complete 1-hour sessions, twice a week for 12 weeks.

Face-to-face physical therapy program (FPT Group) The exercise sessions will take place in a senior center for OAs, lasting 40-60 min, twice a week for 12 weeks; and will include a mixture of cardiovascular, balance, strength, flexibility, and gait exercises.

Regardless of the group, each session will consist of a warm-up activity (5-10 min), main exercise activity (30-40 min), and cool-down activity (5-10 min) following the guidelines of a multicomponent exercise program. Exercise intensity will be controlled based on the Rating of Perceived Exertion (RPE) on the Borg scale, and heart rate measured with a smartwatch before, during and, after each exercise session according to the guidelines of the American College of Sports Medicine (ACSM), as explained below. The warm-up and cool-down activities will include stretching and walking in place (9≤RPE≤10 and 40<55% maximum Heart rate (HRmax)), while the main exercise activity will consist of strength, resistance exercise, cardiovascular exercises and balance exercises (to avoid falls) performed using dumbbells, color-coded resistance bands (Thera-Band; Hygenic Corp.) and a chair (11<RPE≤15 and 55<70 HRmax).

To ensure safety and compliance, exercise training will be supervised by a health professional (physical therapy) who has been appropriately trained (research support stuff). This health professional will provide one-on-one instructions to each participant, according to the target RPE and HRmax (measured with a smartwatch) for each session. All participants will interact with the same health professional.

Specifically in each session, the resistance exercise will be carried out through squats, dumbbells or sitting on the chair using color band (as an example of the exercise progression: yellow (Level 1) band during Weeks 1-4, red (Level 2) band during Weeks 5-8, and green (Level 3) band during Weeks 9-12). This routine, will focus on the main muscle groups in the shoulders, arms, thighs, hips, and calves, included three or four sets with 8-15 repetitions per set. The balance exercise will include two-legged standing, tandem standing, single-legged standing, semi-tandem standing, tandem walking, turning in a circle around the chair, and exercises such as standing on toes, which will focus on postural muscle groups. Cardiovascular exercise will consist of walking at a pace that participants can maintain a continuous conversation at, but that requires some effort. The walk time may increase as the sessions go by (8-15 minutes). The total exercise time was progressively increased from 40-60 minutes over the course of the intervention period. Previous Concurso de Proyectos de Iniciación en Investigación 2024 international studies that analyze synchronous telerehabilitation programs, have used similar exercise protocols.

In the event of an adverse event involving a participant in the FTP group, the AOC 1.1 protocol "Alert system and organization in the event of an emergency" will be used. The participant is assisted and accompanied until the arrival of the emergency medical care service (SAMU). At the same time, other research support personnel will phone a family member. Follow up will then be done.

In the case of a STR group participant, who presents an adverse event, an immediate telephone call will be made to the emergency service and to a registered family member. In addition, communication with the affected user will be always maintained, until the arrival of a family member and/or emergency service. After the event occurs, follow-up will be carried out.

Outcome measures Physical fitness, functional status and quality of life will be examined before and after the interventions. All measurements will be performed by a health professional (technical stuff will be trained) blinded to the group allocation scheme, which will guarantee an unbiassed procedure. Additionally, all measurements will be carried out in a face-to-face meeting and obtained individually, in a place with optimal conditions of privacy, temperature and humidity (a care center to older adults that collaborates with the project). The main outcome for this trial will be lower body strength (evaluated in the 30 second chair stand test) and cardiorespiratory fitness (evaluated using the 2-minutes step test). Secondary outcomes included upper limb strength, dynamic balance, static balance, number of daily steps, functional status, and quality of life.

Physical fitness:

* Lower limb strength will be measured using a five-repetition sit-to-stand test. The OAs will be asked to stand up and sit down, as quickly as possible, five times, from a chair without armrests located on a wall. The time will be measured from the beginning of the movement until the OA manages to stand up for the fifth time. The older adult's arms should be crossed over the chest during the test. The time will be recorded in seconds, and tenths of a second.
* Upper limb strength will be estimated by the grip Strength Test using a previously calibrated BASELINE® brand hydraulic dynamometer. This evaluation will be carried out with the OA seated on a chair with a backrest, shoulders adducted, elbow flexed at 90º, forearm and wrist in a neutral position. The evaluated arm should not rest on any surface and the dynamometer used in a vertical position. OAs will be asked to perform a maximum grip force with their dominant hand for 3 seconds, resting for 1 minute between each repetition, making two attempts. The highest grip value of the repetitions will be used. This protocol is described in ENS 2016-2017.
* Cardiorespiratory fitness will be measured by a 2-minutes step test: The evaluator will count the number of full steps completed by the participant in 2 minutes. A full step is defined as a step performed while raising the knee up to a height corresponding to the midpoint between the patella and the iliac crest.
* Dynamic balance will be measured with the timed up and go test. The OA will be seated on a chair without armrests, with the back against the backrest and feet touching the ground. The OA will be asked to stand up and walk as usual, to a cone located 3 meters away, turn around and return to sit down. This test controls the time it takes to complete the circuit, starting from the moment the OA lifts his/her back from the chair, and ending when returning to the start position. The scale is, normal ≤10 seconds; slight risk of falling 11-20 seconds and, high risk >20 seconds.
* Static balance will be measured using the unipodal stance test. The participant will be asked to cross their arms over their chest, rest their hands on their shoulders, and triple-flex one leg at 90°, staying as long as possible on one foot (maximum of 30 seconds). The test will be repeated three times, the best time obtained will be considered for the study. According to national studies, it is assumed that an OA has a high risk of falling due to not being able to maintain this position for ≥5 seconds.
* Number of daily steps Each participant will wear a digital pedometer for seven days in a row. The steps recorded during the entire time will be added and divided by the number of days of compliance Concurso de Proyectos de Iniciación en Investigación 2024 to obtain the average number of steps per day. Each participant will receive instructions and an illustrative guide with the specific care of the equipment. The classification proposed by Tudor-Locke and Bassett will be used, which indicates that, a number of steps represents the level of physical activity:<2,500 steps/day (basal activity); 2,500 - 4,999 steps/day (limited activity); 5,000-7,499 steps/day (low activity); 7,500-9,999 steps/day (mildly active); 10,000- 12,499 steps/day (active); >12,500 steps/day (highly active).

Functional status:

It will be measured by using the Functional Independence Measure (FIM). It is composed of 18 items, with a total score ranging from 18 to 126, and it allows quantifying the demand for help from third parties that a person needs to perform their daily life activities. The evaluated items include activities of self-care, sphincter control, locomotion, mobility/transfer, and social cognition. For each evaluated activity, the score ranges from 1 - totally dependent, to 7 - totally independent. The FIM is one of the most widely used instruments to carry out functional evaluation in rehabilitation, validated for the elderly, presents clinical validity, agreement between evaluators, test-retest and intra-observer reliability and has been widely used in Chile.

Quality of life:

The Short Form-36 Health Survey in its Spanish version will be used to assess quality of life. The Short Form-36 Health Survey is a self-report instrument that contains 36 questions from 8 dimensions related to people's health: physical function, physical role, bodily pain, vitality, social function, emotional role, mental health, and general health. The score obtained corresponds to values on a scale of 0 to 100. A higher score reflects a better quality of life.

The sociodemographic background of the older adults will be recorded as age, gender (male/female) and geographical origin (rural or urban), educational level (basic <8 years, middle 8-12 years, or higher education >12 years), presence of comorbidities (diabetes mellitus, arterial hypertension, dyslipidemia). Nutritional status will be classified based on the body mass index (BMI). Weight (kg) and height (m) will be combined to report BMI in kg/m^2. Cut-off points will be considered (low weight: <22.9 kg/m2; normal weight: 23.0-27.9 kg/m2; overweight: 28.0-31.9 kg/m2; and obesity: ≥32.0 kg/m2). The questions and the classification indicated in the National Health Survey 2016-2017, will be used.

Statistical analysis Data will be analyzed using SPSS software (version 26 for Windows, IBM, New York, USA). Missing data will be handled by intention-to-treat analysis (multiple imputation method). The description will be made as measures of central tendency and dispersion (continuous variables) and as percentages (categorical variables). Using the Shapiro-Wilk test, the normality of the data will be verified, and a two-step approach for transforming will be applied to the non-normal variables. Homoscedasticity will be analyzed using Levene's test. A 2-way repeated measures analysis of variance (ANOVA) will be used to determine the effects of interventions. The effects of the model are the group (GE; GC), the times (Pretest; Posttest) and their interaction over time (Time x Group). The Bonferroni post hoc test will be applied to identify statistically significant comparisons. The TE will be determined using Cohen's d (<0.2 insignificant; ≥0.2 and ≤0.49 small; ≥0.5 and ≤0.79 moderate; ≥0.8 large). All analyzes will be performed with SPSS v.25 (SPSS, Inc., Chicago, IL, USA) considering p<0.05 and GraphPad Prism v8.

Expected results It is expected that a synchronous telerehabilitation program and a face-to-face physical therapy program improve the main outcome (lower body strength cardiorespiratory fitness) and secondary outcomes (upper limb strength, dynamic balance, static balance, number of steps, functional status, and quality of life) of frail older people. Besides, it is expected that a synchronous telerehabilitation program compared to a face-to-face physical therapy program has equal or greater improvement in the main outcome (lower body strength cardiorespiratory fitness) and secondary outcomes (upper limb strength, dynamic balance, static balance, number of steps, functional status and quality of life) of frail older people. The synchronous telerehabilitation can be a simple, low-cost, and fun alternative to traditional exercise programs to promote active ageing.

ELIGIBILITY:
Inclusion Criteria:

(i) both sexes aged ≥60 years, (ii) community-dwelling older adults, (iii) older adults having frailty according to the modified Fried phenotype scale, (iv) ability to stand up and walk ≥10 meters without assistance technique, (v) Abbreviated Mini Mental State (MMSE) >13 points, (vi) no medical contraindication for physical exercise. In addition, older adults must have a smartphone or tablet, and Internet connection at home. Computer or Internet literacy is not required as an eligibility criterion.

Exclusion Criteria: Those older adults presenting fractures and recent acute myocardial infarction, associated cardiovascular pathology, severe acute respiratory failure, high blood pressure, uncontrolled diabetes mellitus, limitations following instructions, as well as people participating in other exercise program during the project.

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 58 (Estimated)
Dates: Start 2025-04-01 (Estimated); Primary Completion 2025-05-30 (Estimated); Study Completion 2025-08-30 (Estimated)

PRIMARY OUTCOMES:
Lower limb strength | Both groups will be face-to-face assessed one week before and after the 12-week intervention.
  Will be measured using a five-repetition sit-to-stand test. The OAs will be asked to stand up and sit down, as quickly as possible, five times, from a chair without armrests located on a wall. The time will be measured from the beginning of the movement until the OA manages to stand up for the fifth time. The older adult's arms should be crossed over the chest during the test. The time will be recorded in seconds, and tenths of a second.
Cardiorespiratory fitness | Both groups will be face-to-face assessed one week before and after the 12-week intervention.
  Will be measured by a 2-minutes step test: The evaluator will count the number of full steps completed by the participant in 2 minutes. A full step is defined as a step performed while raising the knee up to a height corresponding to the midpoint between the patella and the iliac crest.

SECONDARY OUTCOMES:
Upper limb strength | Both groups will be face-to-face assessed one week before and after the 12-week intervention.
  Will be estimated by the grip Strength Test using a previously calibrated BASELINE® brand hydraulic dynamometer. This evaluation will be carried out with the older people seated on a chair with a backrest, shoulders adducted, elbow flexed at 90º, forearm and wrist in a neutral position. The evaluated arm should not rest on any surface and the dynamometer used in a vertical position. older people will be asked to perform a maximum grip force with their dominant hand for 3 seconds, resting for 1 minute between each repetition, making two attempts. The highest grip value of the repetitions will be used. This protocol is described in Chilean national health survey 2016-2017.
Dynamic balance | Both groups will be face-to-face assessed one week before and after the 12-week intervention.
  Will be measured with the timed up and go test. The older people will be seated on a chair without armrests, with the back against the backrest and feet touching the ground. The older people will be asked to stand up and walk as usual, to a cone located 3 meters away, turn around and return to sit down. This test controls the time it takes to complete the circuit, starting from the moment the older people lifts his/her back from the chair, and ending when returning to the start position. The scale is, normal ≤10 seconds; slight risk of falling 11-20 seconds and, high risk >20 seconds
Static balance | Both groups will be face-to-face assessed one week before and after the 12-week intervention.
  Will be measured using the unipodal stance test. The participant will be asked to cross their arms over their chest, rest their hands on their shoulders, and triple-flex one leg at 90°, staying as long as possible on one foot (maximum of 30 seconds). The test will be repeated three times, the best time obtained will be considered for the study. According to national studies, it is assumed that an older people has a high risk of falling due to not being able to maintain this position for ≥5 seconds
Quality of life | Both groups will be face-to-face assessed one week before and after the 12-week intervention.
  To assess the quality of life, we will use the Short Form-36 Health Survey, Spanish version. The Short Form-36 Health Survey is a self-report instrument that contains 36 questions from 8 dimensions related to people's health: physical function, physical role, bodily pain, vitality, social function, emotional role, mental health, and general health. The score obtained corresponds to values on a scale of 0 to 100. A higher score reflects a better quality of life.
Functional status | Both groups will be face-to-face assessed one week before and after the 12-week intervention.
  It will be measured by using the Functional Independence Measure (FIM). This questionnaire allows quantifying the demand for help from third parties that a person needs to perform their daily life activities. It is composed of 18 items, with a total score ranging from minimum of 18 to a maximum of 126 points. Higher scores reflect a higher level of independence. The evaluated items include activities of self-care, sphincter control, locomotion, mobility/transfer, and social cognition. For each evaluated activity, the score ranges from 1 - totally dependent, to 7 - totally independent. The FIM is one of the most widely used instruments to carry out functional evaluation in rehabilitation, validated for the elderly, presents clinical validity, agreement between evaluators, test-retest and intra-observer reliability and has been widely used in Chile.
Number of daily steps | Both groups will be face-to-face assessed one week before and after the 12-week intervention.
  Each participant will wear a digital pedometer for seven days in a row. The steps recorded during the entire time will be added and divided by the number of days of compliance Concurso de Proyectos de Iniciación en Investigación 2024 to obtain the average number of steps per day. Each participant will receive instructions and an illustrative guide with the specific care of the equipment. We will use the classification proposed by Tudor-Locke and Bassett, which indicates that, a number of steps represents the level of physical activity:<2,500 steps/day (basal activity); 2,500 - 4,999 steps/day (limited activity); 5,000-7,499 steps/day (low activity); 7,500-9,999 steps/day (mildly active); 10,000- 12,499 steps/day (active); >12,500 steps/day (highly active).

OTHER OUTCOMES:
Sociodemographic background | Both groups will be assessed in person one week prior to the 12-week intervention.
  The sociodemographic background of the older adults will be recorded as age, gender (male/female) and geographical origin (rural or urban), educational level (basic <8 years, middle 8-12 years, or higher education >12 years), presence of comorbidities (diabetes mellitus, arterial hypertension, dyslipidemia). Nutritional status will be classified based on the body mass index (BMI). Weight (kg) and height (m) will be combined to report BMI in kg/m^2. Cut-off points will be considered (low weight: <22.9 kg/m2; normal weight: 23.0-27.9 kg/m2; overweight: 28.0-31.9 kg/m2; and obesity: ≥32.0 kg/m2). The questions and the classification indicated in the National Health Survey 2016-2017, will be used.

CONTACTS AND LOCATIONS:
Locations (1):
- Universidad Católica Silva Henríquez, Santiago, Santiago Metropolitan, Chile

REFERENCES:
- [Background] Cramer SC, Dodakian L, Le V, See J, Augsburger R, McKenzie A, Zhou RJ, Chiu NL, Heckhausen J, Cassidy JM, Scacchi W, Smith MT, Barrett AM, Knutson J, Edwards D, Putrino D, Agrawal K, Ngo K, Roth EJ, Tirschwell DL, Woodbury ML, Zafonte R, Zhao W, Spilker J, Wolf SL, Broderick JP, Janis S; National Institutes of Health StrokeNet Telerehab Investigators. Efficacy of Home-Based Telerehabilitation vs In-Clinic Therapy for Adults After Stroke: A Randomized Clinical Trial. JAMA Neurol. 2019 Sep 1;76(9):1079-1087. doi: 10.1001/jamaneurol.2019.1604. PMID 31233135
- [Background] Neo JH, Teo ST, Lee CL, Cai CC. Telerehabilitation in the Treatment of Frozen Shoulder: A Case Report. Int J Telerehabil. 2019 Dec 12;11(2):3-8. doi: 10.5195/ijt.2019.6288. eCollection 2019. PMID 35949924
- [Background] Turolla A, Rossettini G, Viceconti A, Palese A, Geri T. Musculoskeletal Physical Therapy During the COVID-19 Pandemic: Is Telerehabilitation the Answer? Phys Ther. 2020 Aug 12;100(8):1260-1264. doi: 10.1093/ptj/pzaa093. No abstract available. PMID 32386218
- [Background] Velayati F, Ayatollahi H, Hemmat M. A Systematic Review of the Effectiveness of Telerehabilitation Interventions for Therapeutic Purposes in the Elderly. Methods Inf Med. 2020 May;59(2-03):104-109. doi: 10.1055/s-0040-1713398. Epub 2020 Jul 6. PMID 32629502
- [Background] Changizi M, Kaveh MH. Effectiveness of the mHealth technology in improvement of healthy behaviors in an elderly population-a systematic review. Mhealth. 2017 Nov 27;3:51. doi: 10.21037/mhealth.2017.08.06. eCollection 2017. PMID 29430455
- [Background] Wu G, Keyes LM. Group tele-exercise for improving balance in elders. Telemed J E Health. 2006 Oct;12(5):561-70. doi: 10.1089/tmj.2006.12.561. PMID 17042710
- [Background] Solis-Navarro L, Gismero A, Fernandez-Jane C, Torres-Castro R, Sola-Madurell M, Berge C, Perez LM, Ars J, Martin-Borras C, Vilaro J, Sitja-Rabert M. Effectiveness of home-based exercise delivered by digital health in older adults: a systematic review and meta-analysis. Age Ageing. 2022 Nov 2;51(11):afac243. doi: 10.1093/ageing/afac243. PMID 36346736
- [Background] Yuen J, Thiyagarajan CA, Belci M. Patient experience survey in telemedicine for spinal cord injury patients. Spinal Cord. 2015 Apr;53(4):320-3. doi: 10.1038/sc.2014.247. Epub 2015 Jan 27. PMID 25622730
- [Background] Levy CE, Silverman E, Jia H, Geiss M, Omura D. Effects of physical therapy delivery via home video telerehabilitation on functional and health-related quality of life outcomes. J Rehabil Res Dev. 2015;52(3):361-70. doi: 10.1682/JRRD.2014.10.0239. PMID 26230650
- [Background] Schmeler MR, Schein RM, McCue M, Betz K. Telerehabilitation clinical and vocational applications for assistive technology: research, opportunities, and challenges. Int J Telerehabil. 2009 Sep 4;1(1):59-72. doi: 10.5195/ijt.2009.6014. eCollection 2009 Fall. PMID 25945163
- [Background] Irgens I, Rekand T, Arora M, Liu N, Marshall R, Biering-Sorensen F, Alexander M. Telehealth for people with spinal cord injury: a narrative review. Spinal Cord. 2018 Jul;56(7):643-655. doi: 10.1038/s41393-017-0033-3. Epub 2018 Mar 7. PMID 29515211
- [Background] Theodoros D, Russell T. Telerehabilitation: current perspectives. Stud Health Technol Inform. 2008;131:191-209. PMID 18431862
- [Background] Kairy D, Tousignant M, Leclerc N, Cote AM, Levasseur M, Researchers TT. The patient's perspective of in-home telerehabilitation physiotherapy services following total knee arthroplasty. Int J Environ Res Public Health. 2013 Aug 30;10(9):3998-4011. doi: 10.3390/ijerph10093998. PMID 23999548
- [Derived] Cigarroa I, Reyes-Molina D, Vargas-Rios F, Lopez-Alarcon G, Jara-Aceituno S, Riquelme-Hernandez C, Zapata-Lamana R, Parra-Rizo MA. Effectiveness of Synchronous Telerehabilitation Versus Face-to-Face Physical Therapy in Older Adults Who Are Frail: Protocol for a Randomized Controlled Trial. JMIR Res Protoc. 2025 Sep 16;14:e72318. doi: 10.2196/72318. PMID 40957013